CLINICAL TRIAL: NCT02235077
Title: Aldosterone Targeted Neurohormonal Combined With Natriuresis Therapy - HF (ATHENA-HF)
Brief Title: Study of High-dose Spironolactone vs. Placebo Therapy in Acute Heart Failure
Acronym: ATHENA-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00057090; 5U01HL084904 (NIH)
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Heart Diseases; Cardiovascular Diseases; Spironolactone; Aldactone
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Active Comparator): Spironolactone 25mg or 100 mg orally, once daily while in the hospital for 96 hours
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo 25mg or 100mg orally, once daily while in the hospital for 96 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Patients receiving no MRA at home will receive spironolactone 100 mg (4x25 mg capsules) once daily for 96 hours.
  Patients already receiving low-dose MRA at home will be randomized to receive spironolactone 25 mg (1x25 mg capsules) or 100 mg (4x25 mg capsules) in hospital for 96 hours. The patients who are randomized to 25 mg spironolactone will also receive 75 mg placebo (3x25 mg capsules) in order to maintain blinding.
  Other Names: aldactone
  Arms: Spironolactone
Drug: Placebo — Patients receiving no MRA at home will receive 100 mg placebo (4x25 mg capsules) once daily for 96 hours.
  Patients who are randomized to 25 mg spironolactone will also receive 75 mg placebo (3x25 mg capsules) in order to maintain blinding.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to test the hypothesis that high-dose spironolactone will lead to greater proportional reduction in NT-proBNP levels from randomization to 96 hours over standard of care.

DETAILED DESCRIPTION:
Mineralocorticoid receptor antagonist (MRA) therapy is recommended in stable chronic systolic heart failure (HF) and post-infarction HF patients for improving morbidity and mortality. MRA therapy in AHF and in high doses is less well studied. The effectiveness and safety of early high dose MRA therapy in AHF is supported by a single-blind study showing lower risk of worsening renal function and need for loop diuretics, and improved congestion. MRA therapy in AHF may improve outcomes by relieving congestion at higher doses through their natriuretic property, in addition to preventing the deleterious effects of exacerbation of neuro-hormonal activation by loop diuretics.

This randomized, double blind, placebo-controlled study of high-dose spironolactone vs. placebo (for patients not receiving MRA at home) or low-dose spironolactone (for patients already receiving low-dose spironolactone) in AHF, will enroll 360 participants at approximately 30 clinical centers. After obtaining informed consent, subjects who fulfill all the inclusion criteria and none of the exclusion criteria will be randomized. Randomization will be performed by using procedures determined by the Coordinating Center (CC).

* Patients receiving no MRA therapy at baseline will be randomized to receive either spironolactone 100 mg or placebo daily for 96 hours.
* Patients already receiving low-dose spironolactone at baseline (12.5 mg or 25 mg daily) will be randomized to 100 mg or 25 mg spironolactone daily for 96 hours.

Within 24 hours prior to randomization, all study participants will undergo:

* Medical History
* Review of medications including pre-hospital loop diuretics, MRA, and potassium doses
* Physical examination, vital signs and body weight
* Measurement of creatinine, blood urea nitrogen (BUN), and electrolytes
* Dyspnea Relief Assessments (7-point Likert and Visual Analog Scale)
* Serum pregnancy test for all women of childbearing potential
* Collection of samples for measurement of NT-proBNP levels (Core Lab)

Study drug will be initiated as follows:

* Patients receiving no MRA therapy at baseline: 4x25 mg study capsules once daily; starting dose 100 mg spironolactone or placebo; if dose adjustment is required, active capsules will be adjusted by pharmacy to achieve the required dose.
* Patients already receiving low-dose spironolactone at baseline: 4x25 mg study capsules once daily; one capsule containing 25 mg spironolactone and 3x25 mg study capsules containing spironolactone or placebo; if dose adjustment is required, active capsules will be adjusted by pharmacy to achieve the required dose.

Patients will be followed every 24 hours following randomization through 96 hours. Study drug will be administered daily for 96 hours. Study drug administration time is anchored to time of randomization. Dose adjustments (continue, hold, stop) are permitted according to serum K+ and renal function.

Assessment at 24 hours post randomization includes: Review of medications, body weight, fluid intake/urine output, creatinine, blood urea nitrogen (BUN), and electrolytes, and adverse events.

If the 24 hour assessment is also the day of discharge, include:

* Physical exam / Vital signs
* Dyspnea Relief (7-Point Likert and VAS) worksheets
* Biomarkers (NT-proBNP) (Core Lab)

Assessment at 48 hours post randomization includes: Review of medications, physical exam/vital signs, body weight, fluid intake/urine output, Dyspnea Relief (7-Point Likert and VAS) worksheets, creatinine, blood urea nitrogen (BUN), and electrolytes, biomarker levels (NT-proBNP) by Core Lab.

Assessment at 72 hours post randomization includes: Review of medications, body weight, fluid intake/urine output, creatinine, blood urea nitrogen (BUN), and electrolytes, and adverse events.

If the 72 hour assessment is also the day of discharge, include:

* Physical exam / Vital signs
* Dyspnea Relief (7-Point Likert and VAS) worksheets
* Biomarkers (NT-proBNP) (Core Lab)

Assessment at 96 hours post randomization includes: Review of medications, physical exam/vital signs, body weight, fluid intake/urine output, creatinine, blood urea nitrogen (BUN), and electrolytes, Dyspnea Relief (7-Point Likert and VAS), and biomarker levels (NT-proBNP) by Core Lab.

If patient is clinically euvolemic in less than 96 hours, the investigator may consider changing loop diuretics to oral dose.

Study drug will be discontinued after 96 hours and further use of MRA will be left to the treating physician's discretion.

Assessment at Discharge: If discharge occurs after the 96 hour assessment but prior to the 30 day follow-up telephone call,the following will be documented: Medication review (prescribed medications at the time of discharge), body weight (if available), creatinine, blood urea nitrogen (BUN), and electrolytes (if available), and adverse events.

Ejection fraction data will be obtained from echocardiogram within 6 months prior to randomization. Those patients who do not have an echocardiogram recorded within this time frame will get an echocardiogram, nuclear perfusion study, MRI, or MUGA performed prior to the 96 hour in-hospital assessment to ascertain ejection fraction.

Follow-up Telephone Call at Day 30: All participants will be contacted by telephone at day 30 (+3 days) following randomization to assess tertiary endpoints, including medication use and adverse events.

Follow-up Telephone Call at Day 60: All participants will be contacted by telephone at day 60 (+/-3 days) following randomization to assess vital status.

During the consent process, patients will be asked if interested in donating samples and data for research purposes via a biorepository and/or genetic study. Based on site and IRB preference, this optional part of the study may be incorporated into the main consent or may be a separate consent and IRB application.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥21 years old
* Admitted to hospital for AHF with at least 1 symptom (dyspnea, orthopnea, or fatigue) and 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography) of congestion
* Patient must be randomized within 24 hours of first IV diuretic dose administered for the current episode of decompensation (regardless of where the diuretic was given e.g. office, ED, ambulance, hospital etc.)
* Estimated GFR of ≥30 mL/min/1.73m2 determined by the MDRD equation
* Serum K+ ≤5.0 mmol/L at enrollment
* NT-proBNP ≥1000 pg/mL or BNP ≥250 pg/mL, measured within 24h from randomization
* Not on MRA or on low-dose spironolactone (12.5 mg or 25 mg daily) at baseline

Exclusion Criteria:

* Taking eplerenone or >25 mg spironolactone at baseline
* eGFR < 30 ml/min/1.73m2
* Serum K+ >5.0 mmol/L. If a repeat measurement within the enrollment window is <5.0, the patient can be considered for inclusion.
* Systolic blood pressure <90 mmHg
* Hemodynamically significant arrhythmias or defibrillator shock within 1 week
* Acute coronary syndrome currently suspected or within the past 4 weeks
* Severe liver disease (ALT or AST >3 x normal, alkaline phosphatase or bilirubin >2x normal)
* Active infection (current use of oral or IV antimicrobial agents)
* Active gastrointestinal bleeding
* Active malignancy other than non-melanoma skin cancers
* Current or planned mechanical circulatory support within 30 days
* Post cardiac transplant or listed for transplant and expected to receive one within 30 days
* Current inotrope use
* Complex congenital heart disease
* Primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy, acute myocarditis, constrictive pericarditis or tamponade
* Previous adverse reaction to MRAs
* Enrollment in another randomized clinical trial during index hospitalization

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University Health Systems; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (22):
- United States (22):
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston VA Healtcare System, West Roxbury, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - University Hospitals - Case Medical Center, Cleveland, Ohio
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Michael Debakey VA Medical Center, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Utah VA Medical Center, Salt Lake City, Utah
  - The University of Vermont- Fletcher Allen Health Care, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Greene SJ, Felker GM, Giczewska A, Kalogeropoulos AP, Ambrosy AP, Chakraborty H, DeVore AD, Fudim M, McNulty SE, Mentz RJ, Vaduganathan M, Hernandez AF, Butler J. Spironolactone in Acute Heart Failure Patients With Renal Dysfunction and Risk Factors for Diuretic Resistance: From the ATHENA-HF Trial. Can J Cardiol. 2019 Sep;35(9):1097-1105. doi: 10.1016/j.cjca.2019.01.022. Epub 2019 Feb 7. PMID 31230825
- [Derived] Butler J, Anstrom KJ, Felker GM, Givertz MM, Kalogeropoulos AP, Konstam MA, Mann DL, Margulies KB, McNulty SE, Mentz RJ, Redfield MM, Tang WHW, Whellan DJ, Shah M, Desvigne-Nickens P, Hernandez AF, Braunwald E; National Heart Lung and Blood Institute Heart Failure Clinical Research Network. Efficacy and Safety of Spironolactone in Acute Heart Failure: The ATHENA-HF Randomized Clinical Trial. JAMA Cardiol. 2017 Sep 1;2(9):950-958. doi: 10.1001/jamacardio.2017.2198. PMID 28700781
- [Derived] Butler J, Hernandez AF, Anstrom KJ, Kalogeropoulos A, Redfield MM, Konstam MA, Tang WH, Felker GM, Shah MR, Braunwald E. Rationale and Design of the ATHENA-HF Trial: Aldosterone Targeted Neurohormonal Combined With Natriuresis Therapy in Heart Failure. JACC Heart Fail. 2016 Sep;4(9):726-35. doi: 10.1016/j.jchf.2016.06.003. Epub 2016 Aug 10. PMID 27522631

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone: Spironolactone 25mg or 100 mg orally, once daily while in the hospital for 96 hours
  Spironolactone: Patients receiving no MRA at home will receive either spironolactone 100 mg or matching placebo (4x25 mg study capsules) once daily for 96 hours.
  Patients already receiving low-dose MRA at home will receive spironolactone 100 mg vs. 25 mg (1x25 mg spironolactone and 3 placebo study capsules) in hospital for 96 hours.
- Placebo: Placebo 25mg or 100mg orally, once daily while in the hospital for 96 hours
  Placebo: Patients receiving no MRA at home will receive either spironolactone 100 mg or matching placebo (4x25 mg study capsules) once daily for 96 hours.
  Patients already receiving low-dose MRA at home will receive spironolactone 100 mg vs. 25 mg (1x25 mg spironolactone and 3 placebo study capsules) in hospital for 96 hours.
Period: Overall Study
Arm/Group | Spironolactone | Placebo
Started | 182 | 178
Completed | 164 | 159
Not Completed | 18 | 19
Not completed — Death | 5 | 7
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 182 | 178 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (13.7) | 63.5 (14.4) | 64.7 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 129
  Male | 117 | 114 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 180 | 172 | 352
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 74 | 77 | 151
  White | 101 | 99 | 200
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 96 Hour Change in NT-proBNP
Description: The Core Laboratory at Vermont will determine NT-proBNP levels for calculation of the endpoint from samples obtained at randomization and 96 hours respectively. NT-proBNP was converted to log scale.
Time Frame: Randomization to 96 hours
Measure: Mean (Standard Deviation); unit: log pg/ml
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 182 | 178
log pg/ml | -0.58 (0.69) | -0.61 (0.72)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.5688, Regression, Linear; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.11 to 0.20]

2. Secondary Outcome: 96 Hour Change in Clinical Congestion Score
Description: Clinical congestion score will be assessed at randomization, 96 hours, and at discharge. Scale consisted of sum of six signs and symptoms of congestion, each scored 0-3. Zero indicates no sign/symptom and 3 indicates worst case of sign/symptom. Score range 0-18 with 18 being worst score.
Time Frame: Randomization through 96 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 182 | 178
units on a scale | -5.59 (3.34) | -5.82 (3.32)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.4155, Regression, Linear; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.35 to 0.86]

3. Secondary Outcome: 96 Hour Change in Dyspnea Likert Score
Description: Dyspnea relief via 7-point Likert scale will be assessed at randomization, 96 hours, and at discharge. The Likert score was defined as 1=markedly improved, 2=moderately improved, 3=minimally improved; 4=no change, 5=minimally worse, 6=moderately worse, and 7=markedly worse as compared with the degree of dyspnea present at randomization.
Time Frame: Randomization through 96 hours
Population: All data for completed assessments was analyzed. For outcomes where the number of participants analyzed is less than 182 spironolactone / 178 placebo, the number of subjects analyzed represents the number of subjects for whom the data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 166 | 163
Participants
  Markedly improved | 64 | 79
  Moderately improved | 56 | 39
  Minimally improved | 24 | 18
  No change | 17 | 21
  Minimally worse | 4 | 5
  Moderately worse | 0 | 0
  Markedly worse | 1 | 1
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.3039, Chi-squared; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.83 to 1.81]

4. Secondary Outcome: 96 Hour Change in Serum Creatinine
Description: Renal function via serum creatinine, will be assessed at randomization and daily through 96 hours
Time Frame: Randomization through 96 hours
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 100 | 101
mg/dl | 0.15 (0.30) | 0.16 (0.30)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.7673, Regression, Linear; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.09 to 0.07]

5. Secondary Outcome: 96 Hour Net Fluid Output
Description: Fluid intake and urine output will be assessed daily while in hospital through 96 hours. Net fluid output (output minus input) through 96 hours is reported.
Time Frame: Randomization through 96 hours
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 87 | 96
ml | 5824 (4007) | 5507 (3633)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.5734, Regression, Linear; Mean Difference (Final Values) = 319.2, 95% CI 2-sided [-797.4 to 1435.8]

6. Secondary Outcome: 96 Hour Change in Body Weight
Description: Baseline body weight assessment will be completed, and changes in weight documented daily through 96 hours or earlier discharge
Time Frame: Randomization through 96 hours or earlier discharge
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 182 | 178
pounds | -8.1 (10.7) | -7.5 (9.5)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.3528, Regression, Linear; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-3.05 to 1.01]

7. Secondary Outcome: 96 Hour Change in Serum Potassium Levels
Description: Change in serum potassium levels at 96 hours as compared to baseline.
Time Frame: Baseline, 96 hours
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 99 | 101
mEq/L | 0.31 (0.54) | 0.15 (0.69)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.0846, Regression, Linear; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.02 to 0.25]

8. Secondary Outcome: Change in Loop Diuretics Requirements From Baseline to 30 Days
Description: Medications will be reviewed to assess loop diuretic dose requirements through Day 30 following randomization
Time Frame: Randomization through Day 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 164 | 158
mg | 19.66 (69.95) | 30.70 (68.29)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.0842, Regression, Linear; Mean Difference (Final Values) = -12.17, 95% CI 2-sided [-25.98 to 1.65]

9. Secondary Outcome: Presence of Outpatient Worsening Heart Failure Symptoms Through Day 30
Description: Outpatient worsening heart failure symptoms will be assessed from discharge through Day 30
Time Frame: Hospital discharge through Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 166 | 163
Participants | 19 | 17
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.7628, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.56 to 2.23]

10. Secondary Outcome: 96 Hour Change in Dyspnea Visual Analog Scale
Description: Dyspnea visual analog scale change from randomization to 96 hours. Scale range 0-100 with 100 being the best possible score.
Time Frame: Randomization to 96 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 182 | 178
units on a scale | 17.2 (25.0) | 17.9 (24.6)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.6102, Regression, Linear; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-5.02 to 2.95]

11. Other Pre Specified Outcome: Day 60 Mortality
Description: All participants will be contacted by telephone at 60 days, +/- 3 days post randomization to assess vital status (death).
Time Frame: 60 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 182 | 178
Participants | 8 | 10
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.5818, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.29 to 1.99]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected by the sites from randomization through 30 days, but was not collected on the case report form. Only Serious Adverse Events were collected on the data forms.
Description: Adverse event data was collected by the sites from randomization through 30 days, but was not collected on the case report form.
Arm/Group | Spironolactone | Placebo
All-Cause Mortality (participants affected / at risk) | 5/182 | 7/178
Serious Adverse Events (participants affected / at risk) | 21/182 | 13/178
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=182) | Placebo (N=178)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemmorhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Protalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
H1N1 Influenza (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-procedural haemotoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemotoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1)
Delerium (Psychiatric disorders) | 1 (1) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Bronchial haemmorhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To minimize the probability of inaccurate data in published materials, it is the policy of the Heart Failure Network that all data and text considered for all papers, and all abstracts for presentation at scientific meetings be submitted to the Publication and Presentation Subcommittee, the NHLBI Project Officer, and the Coordinating Center for review and approval prior to presentation or publication.